CLINICAL TRIAL: NCT06011070
Title: Pilot Randomised Trial of a Brief Online Personalised Feedback Intervention for the UK Context Designed to Prevent, Reduce, and Address Gambling Harm
Brief Title: Brief Online Personalised Feedback Intervention for Gambling Harm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HR-22/23-36398
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Problem Gambling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gambling Personalised Feedback (Experimental): The intervention is a brief online intervention designed to provide personalized normative feedback aimed at motivating reductions in gambling
  Interventions: Behavioral: Gambling Personalised Feedback
- Control (No Intervention): No intervention Control

INTERVENTIONS:
Behavioral: Gambling Personalised Feedback — The intervention is a brief online intervention designed to provide personalized normative feedback aimed at motivating reductions in gambling
  Arms: Gambling Personalised Feedback

SUMMARY:
Purpose and significance A brief self-directed online personalised feedback intervention was developed for the UK context designed to prevent, reduce, and address gambling harm. The intervention, which also comes in a paper format, comprises of normative feedback and personalised information on the risk of gambling above lower-risk gambling guidelines. The content is based on recent work adapting the Canadian lower-risk gambling guidelines to the UK context. The purpose of this exploratory research is to conduct the first randomised controlled trial of this intervention. Further, given the increased prevalence of online gambling, the project will target this at-risk population.

Rationale This project will generate participant feedback on the intervention important to improve its utility. The project will also produce publishable findings on the intervention's efficacy. This evaluation provides a necessary first step towards the wide-spread implementation of this free-of-charge intervention in the UK.

Methodology First, using methods developed in our previous research, we will rapidly recruit 926 online gambling participants with moderate or problem gambling from an existing online panel of UK residents. These participants will be randomised to receive the self-directed online intervention or assigned to a no intervention control group. Participants will be followed-up up at one- and three-months to provide detailed feedback on their impressions of the intervention (and what further modifications are needed) and to assess the short-term impact of the intervention on gambling frequency and harm.

Potential implications of the proposed research The intervention can be accessed at any time of the day and allow the delivery of help without requiring face-to-face contact. Online interventions also have the potential to promote reductions in social inequalities through reducing barriers to accessible care. At present, there appears to be no UK online at-risk gambling intervention that is publicly available.

ELIGIBILITY:
Inclusion Criteria:

* Problem gambling severity index score of 3 or more
* Willingness to complete 1 and 3-month follow-up surveys

Exclusion Criteria

* Do not live in the United Kingdom
* Incorrectly answer attention check question on baseline survey
* Do not endorse that they answered all questions truthfully on the baseline survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1586 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
number of days gambled in the last month | 1 and 3 months
  The number of days the participants reports gambling in the past month

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes